CLINICAL TRIAL: NCT00341731
Title: Environmental Factors in the Development of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901047; 01-E-N047
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2008-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Cystic Ovaries; Environmental Factors; Heritability; Hyperandrogenism; Twin Study
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Cysts; Hyperandrogenism

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is manifested as a heterogeneous mixture of clinical and bichemical characteristics that complicate study of its etiology. It is currently unclear to what extent PCOS-associated traits (hyperandrogenism, hyperinsulinemia, insulin resistance, type 2 diabetes, dyslipidemia, hypertension, obesity, and coronary artery disease) are the result of environmental factors or genetic predisposition. We propose to conduct a twin study to investigate the possibility that environmental factors are important in the development of the PCOS phenotype. Twin studies are considered to be the gold standard for determining the extent of heritability of a trait. The proposal described here is only for Step 1 of a larger, multi-step study. The major goal of step 1 is to identify a large cohort of twin pairs, in which at least one member of each pair is likely to have PCOS.

Participants for this study will come from the Mid-Atlantic Twin Registry (MATR). Many (3283) potential participants have already been identified based on their answers to a preliminary MATR screening questionnaire. Out of the approximately 7145 twin women of reproductive age who completed these MATR screening questionnaires, 1803 women reported irregular periods, 954 reported ovarian cysts, and 526 reported both irregular periods and ovarian cysts. Many of the women in this last group are likely to have PCOS. They represent 7.4% of the total sample, matching current estimates of PCOS prevalence (4-7%) in reproductive age women. We will also add new twin pairs who meet the criteria (irregular periods and evidence of PCOS or cystic ovaries) as they are recruited into the MATR and take the preliminary surveys. According to MATR statistics, about 33% of twin pairs are monozygotic (MZ, identical). Therefore, approximately 174 of the 526 women likely to have PCOS are members of a MZ pair.

Step 1 of the proposed study consists of a telephone survey of the 3282 women with irregular periods and/or ovarian cysts. The survey will be conducted by the MATR. The instrument to be used contains a series of simple and direct questions and will take about 10 minutes to complete. The questions were designed to identify PCOS and their content deals with the frequency of menstrual periods (six or fewer per year being a major diagnostic criterion), a previous diagnosis of PCOS, obesity, excess facial hair and other evidence of hyperandrogenism. The women will also be asked if t...

DETAILED DESCRIPTION:
Polycystic Ovary Syndrome (PCOS) is manifested as a heterogeneous mixture of clinical and bichemical characteristics that complicate study of its etiology. It is currently unclear to what extent PCOS-associated traits (hyperandrogenism, hyperinsulinemia, insulin resistance, type 2 diabetes, dyslipidemia, hypertension, obesity, and coronary artery disease) are the result of environmental factors or genetic predisposition. We propose to conduct a twin study to investigate the possibility that environmental factors are important in the development of the PCOS phenotype. Twin studies are considered to be the gold standard for determining the extent of heritability of a trait. The proposal described here is only for Step 1 of a larger, multi-step study. The major goal of step 1 is to identify a large cohort of twin pairs, in which at least one member of each pair is likely to have PCOS.

Participants for this study will come from the Mid-Atlantic Twin Registry (MATR). Many (3283) potential participants have already been identified based on their answers to a preliminary MATR screening questionnaire. Out of the approximately 7145 twin women of reproductive age who completed these MATR screening questionnaires, 1803 women reported irregular periods, 954 reported ovarian cysts, and 526 reported both irregular periods and ovarian cysts. Many of the women in this last group are likely to have PCOS. They represent 7.4% of the total sample, matching current estimates of PCOS prevalence (4-7%) in reproductive age women. We will also add new twin pairs who meet the criteria (irregular periods and evidence of PCOS or cystic ovaries) as they are recruited into the MATR and take the preliminary surveys. According to MATR statistics, about 33% of twin pairs are monozygotic (MZ, identical). Therefore, approximately 174 of the 526 women likely to have PCOS are members of a MZ pair.

Step 1 of the proposed study consists of a telephone survey of the 3282 women with irregular periods and/or ovarian cysts. The survey will be conducted by the MATR. The instrument to be used contains a series of simple and direct questions and will take about 10 minutes to complete. The questions were designed to identify PCOS and their content deals with the frequency of menstrual periods (six or fewer per year being a major diagnostic criterion), a previous diagnosis of PCOS, obesity, excess facial hair and other evidence of hyperandrogenism. The women will also be asked if they have a living twin sister. On the basis of this survey, women will be identified who are likely to have PCOS and have a living female twin.

ELIGIBILITY:
* INCLUSION CRITERIA:

The only criteria for inclusion into this study are that participants be female twins over the age of 18 and of reproductive age.

Participants will not be excluded based on race, ethnicity or religion.

EXCLUSION CRITERIA:

Women under the age of 18 will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia